CLINICAL TRIAL: NCT06090461
Title: A Non-Interventional Study to Generate Real-World Evidence on the Cardiovascular Safety of CONTRAVE® in the United States (U.S.)
Brief Title: Real-World Evidence on the Cardiovascular Safety of CONTRAVE® in the United States (U.S.)
Acronym: HOA
Status: Completed | Type: Observational
Sponsor: Currax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Cardiovascular Safety Study
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Contrave/Mysimba: A fixed-dose combination of 8 milligrams (mg) of naltrexone hydrochloride (HCl) (an opioid receptor antagonist), and 90 mg of bupropion HCl (a selective neuronal re-uptake inhibitor of noradrenaline and dopamine), delivered through extended-release oral tablets.
- Lorcaserin: A total of one 10 mg tablet administered orally twice daily; or one 20 mg tablet administered orally once daily. Lorcaserin was included as an active comparator to reduce bias.
- Naltrexone and Bupropion (N&B): N&B concomitant use, ultimately as a proxy for initiation, was defined as a record for naltrexone followed by initiation of bupropion, or bupropion followed by initiation of naltrexone, within 15 days of each other.

SUMMARY:
The fixed-dose combination of naltrexone 8mg and bupropion 90mg extended-release oral tablet is marketed under the trade name CONTRAVE® in the U.S. In this protocol, the investigators propose to generate real-world evidence (RWE) from electronic health records (EHR) and linked claims data to assess the cardiovascular safety of CONTRAVE® and all combined use of naltrexone and bupropion (NB) in usual clinical practice.

DETAILED DESCRIPTION:
The study will assess whether patients who initiate treatment with NB are at an elevated risk of MACE compared with patients who initiated treatment with lorcaserin, an active comparator chosen to reduce potential confounding.

The cohorts for all study objectives will be drawn from a large electronic health records (EHR) data source, representing a geographically diverse patient population. The data will include diagnoses, procedures, medications (prescribed and administered), clinical measures (biometric and laboratory values), and observations derived from clinical notes. A subset of the population will have linked, adjudicated claims data available to support sensitivity analyses.

The study's main objective is to compare the incidence of the primary endpoint (MACE) between initiators of NB and initiators of lorcaserin. The study will also compare the incidence of the secondary endpoint, consisting of each component of MACE, between initiators of NB and initiators of lorcaserin, across the following subgroups: Patients with obesity (i.e., most recent BMI measurement ≥30 kg/m2); Patients with a diagnosis of hypertension, regardless of BMI; Patients with a diagnosis of type 2 diabetes mellitus, regardless of BMI; Patients with a diagnosis of dyslipidemia, regardless of BMI.

The study's additional objectives aimed at testing the robustness of the methods are:

To assess the comparability of findings from an EHR study to those of a 2018 clinical trial, aligning with the Randomized Control Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT DUPLICATE) Initiative; To quantify differences in cardiovascular safety endpoints between the clinical trial and the results of this EHR study; To conduct other sensitivity analyses, including a self-controlled, case-crossover analysis to quantify the potential effect of NB on MACE.

ELIGIBILITY:
For the main objective (1.0, 1.1), patients are eligible if they meet the following Inclusion Criteria:

* Have at least one prescription for NB between September 2014 and February 2020, including concurrent prescriptions (within 15 days) for naltrexone and bupropion; or have at least one prescription for lorcaserin;
* Have at least 180 days of data available prior to cohort entry with no evidence of prescriptions or dispensings of NB or lorcaserin;
* Have at least one BMI value available in the 180 days prior to cohort entry, inclusive of the index date;
* Have documentation of at least one outpatient medical visit 180 or more days prior to cohort entry, and at least one healthcare interaction in the 180 days prior to cohort entry;
* Are at least 18 years of age on the cohort entry date.

For the main objective, patients are not eligible if they have a diagnosis of any of the following conditions in the 180 days before the cohort entry date:

* Epilepsy;
* Bulimia;
* Anorexia nervosa;
* Surgical procedure for weight loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary study population includes initiators of NB or the active comparator, lorcaserin.
Sampling Method: Non-Probability Sample
Enrollment: 31889 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Currax Pharmaceuticals, Brentwood, Tennessee, United States

REFERENCES:
- [Result] Kyle M, Burns D, Murray CR, Watson H, Swaney J, Spevack S, Leonhard M, Simon M, Moynihan E, Lapane KL, Wang SV, Longo CL, Ritchey ME, Dore DD. Cardiovascular safety of fixed-dose extended-release naltrexone/bupropion in clinical practice. Obes Pillars. 2025 Feb 17;13:100169. doi: 10.1016/j.obpill.2025.100169. eCollection 2025 Mar. PMID 40104005

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrave/Mysimba | Lorcaserin | Naltrexone and Bupropion (N&B)
Started | 12475 | 12171 | 7243
Completed | 12475 | 12171 | 7243
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contrave/Mysimba | Lorcaserin | Naltrexone and Bupropion (N&B) | Total
Number analyzed (Participants) | 12475 | 12171 | 7243 | 31889
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 47.6 (11.9) | 48.1 (12.2) | 45.5 (13.4) | 47.1 (1.38)
Sex/Gender, Customized [Number; unit: Percentage]
  Female | 82.3 | 81.8 | 65.6 | 77
  Male | 17.7 | 18.2 | 34.4 | 23
Race/Ethnicity, Customized [Number; unit: Percentage of participants]
  Hispanic/Latino | 6.3 | 7.2 | 5.9 | 6
  Not Hispanic/Latino | 68.3 | 69.2 | 65.7 | 68
  Unknown | 25.3 | 23.5 | 28.3 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Major Adverse Cardiovascular Events (MACE) Between Initiators of CONTRAVE®/MYSIMBA® or N&B and Initiators of Lorcaserin.
Description: The primary study endpoint is MACE, defined as the composite of:
  * Medically attended non-fatal acute myocardial infarction (AMI);
  * Medically attended non-fatal stroke;
  * Cardiovascular death.
Time Frame: Up to 113 months
Measure: Number; unit: Events
Arm/Group | Contrave/Mysimba | Lorcaserin | Naltrexone and Bupropion (N&B)
Number analyzed (Participants) | 12475 | 12171 | 7243
Events
  AMI | 26 | 36 | 10
  Stroke | 6 | 5 | 5
  Death | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 113 months
Description: For this study using previously collected and deidentified electronic healthcare data, the research team did not anticipate any new adverse events to be identified.
Arm/Group | Contrave/Mysimba | Lorcaserin | Naltrexone and Bupropion (N&B)
All-Cause Mortality (participants affected / at risk) | 0/12475 | 0/12171 | 1/7243
Serious Adverse Events (participants affected / at risk) | 63/12475 | 81/12171 | 31/7243
Other Adverse Events (participants affected / at risk) | 0/12475 | 0/12171 | 0/7243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contrave/Mysimba (N=12475) | Lorcaserin (N=12171) | Naltrexone and Bupropion (N&B) (N=7243)
AMI (Cardiac disorders) | 26 | 36 | 10
Stroke (Cardiac disorders) | 6 | 5 | 5
MACE (Cardiac disorders) | 31 | 40 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT06090461/Prot_SAP_000.pdf